CLINICAL TRIAL: NCT02252068
Title: Behavioral Treatment Development for Co-occurring Opioid Dependence and Anxiety Disorders
Brief Title: Study of Treatment for Opioid Dependence and Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, McHugh, R. Kathryn, Associate Psychologist, Division of Alcohol and Drug Abuse, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23DA035297 (NIH)
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Anxiety Disorders; Opiate Addiction
MeSH Terms: conditions — Anxiety Disorders; Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- I-CBT feasibility pilot (Other): Open trial of I-CBT
  Interventions: Behavioral: I-CBT
- I-CBT randomized trial (Experimental): I-CBT in randomized trial.
  Interventions: Behavioral: I-CBT
- IDC randomized trial (Active Comparator): Comparison condition (Individualized Drug Counseling) in randomized trial.
  Interventions: Behavioral: IDC

INTERVENTIONS:
Behavioral: I-CBT — New cognitive behavioral therapy treatment manual developed to treat co-occurring anxiety and opioid dependency disorders.
  Arms: I-CBT feasibility pilot; I-CBT randomized trial
Behavioral: IDC — Individual Drug Counseling manual that has demonstrated efficacy for the treatment of drug dependence.
  Arms: IDC randomized trial

SUMMARY:
Anxiety is highly prevalent among individuals with opioid dependence and confers greater risk for continued opioid use and poor treatment outcomes. However, there are currently no efficacious treatments available for co-occurring opioid dependence and anxiety. The ultimate aims of this trial are the development and testing of a novel integrated cognitive behavioral treatment (I-CBT) for co-occurring opioid dependence and anxiety disorders. This clinical trial consists of two phases: (1) open-trial pilot (2) randomized control trial. We hypothesize that I-CBT will be a feasible and acceptable treatment that will result in significant reductions in anxiety and opioid use.

DETAILED DESCRIPTION:
This Stage 1 behavioral treatment development trial involves two stages: manual development and pilot testing in an open trial, and a small randomized controlled trial. In both phases, opioid use and anxiety symptoms will be measured as the primary clinical outcome, along with measures of feasibility and patient satisfaction. These results will be used to further refine the treatment manual and to evaluate whether this treatment may enhance outcomes for adults with co-occurring opioid dependence and anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* meet current Diagnostic and Statistical Manual of Mental Disorders 5th edition diagnostic criteria for opioid use disorder
* currently prescribed pharmacotherapy for opioid dependence
* have used opioids illicitly within the previous 90 days
* clinically-significant anxiety
* meet current diagnostic criteria for a Diagnostic and Statistical Manual of Mental Disorders 5th edition anxiety disorder
* able to read and provide informed consent
* intend to remain in the geographical area for the duration of the study period

Exclusion Criteria:

* meet criteria for a current substance use or psychiatric disorder requiring a level of care higher than outpatient
* currently receiving cognitive behavioral therapy
* recent initiation of a psychiatric medication, defined as less than 4 weeks on a stable dose; not including PRN medications for sleep
* are receiving and taking an as-needed (PRN) prescription for benzodiazepines
* presence of a psychiatric or medical condition that would interfere with participation or that requires additional care (e.g. psychosis, acute suicidality)
* were admitted to McLean Hospital for their current treatment episode on an involuntary status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-01; Primary Completion 2019-10-24 (Actual); Study Completion 2019-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca K McHugh, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the randomized controlled trial, 6 participants completed a baseline assessment but dropped out prior to randomization.
Groups:
- RCT I-CBT: Randomized controlled trial: Integrated Cognitive-Behavioral Therapy Arm
  I-CBT: New cognitive behavioral therapy treatment manual developed to treat co-occurring anxiety and opioid dependency disorders.
- RCT IDC: Randomized Controlled Trial: Individual Drug Counseling Arm
  IDC: Individual Drug Counseling manual that has demonstrated efficacy for the treatment of drug dependence.
Period: Overall Study
Arm/Group | I-CBT Feasibility Pilot | RCT I-CBT | RCT IDC
Started | 5 | 13 | 13
Completed | 3 | 13 | 13
Not Completed | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- I-CBT RCT: Randomized control trial of I-CBT vs ICD
  I-CBT: New cognitive behavioral therapy treatment manual developed to treat co-occurring anxiety and opioid dependency disorders.
- IDC RCT: Randomized control trial of I-CBT vs ICD
  IDC: Individual Drug Counseling manual that has demonstrated efficacy for the treatment of drug dependence.
- Total: Total of all reporting groups
Arm/Group | I-CBT Feasibility Pilot | I-CBT RCT | IDC RCT | Total
Number analyzed (Participants) | 5 | 13 | 13 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (8.3) | 33.9 (10.5) | 31.8 (9.6) | 32.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 3 | 8
  Male | 4 | 9 | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 12 | 13 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 13 | 13 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 13 | 13 | 31

OUTCOME MEASURES:

1. Primary Outcome: Urine-confirmed Self-reported Weeks of Opioid Use
Description: Number of weeks of opioid use at Week 12 for the last 4 weeks of treatment (Weeks 9-12), as assessed by self-report and validated by urine drug screen
Time Frame: Week 12
Population: Due to partial missing data, the analysis population does not reflect the full sample. Specifically, missing data for 2 participants in RCT: I-CBT arm.
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- RCT: I-CBT: Randomized control trial of I-CBT vs ICD
  I-CBT: New cognitive behavioral therapy treatment manual developed to treat co-occurring anxiety and opioid dependency disorders.
- RCT IDC: Randomized control trial of I-CBT vs ICD
  IDC: Individual Drug Counseling manual that has demonstrated efficacy for the treatment of drug dependence.
Arm/Group | I-CBT Feasibility Pilot | RCT: I-CBT | RCT IDC
Number analyzed (Participants) | 3 | 11 | 13
weeks | 1 (1.73) | .36 (1.2) | .31 (.85)

2. Primary Outcome: Anxiety Symptom Severity
Description: Hamilton Anxiety Rating Scale (HADS) score. Measure assesses the severity of anxiety symptoms. Total scale scores are reported. Higher scores reflect worse outcome. The range of possible scores is 0-56.
Time Frame: Week 12
Population: Due to partial missing data, not all participants are included in this analysis. Specifically, missing data for 1 participant in the RCT: I-CBT arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | I-CBT Feasibility Pilot | RCT: I-CBT | RCT IDC
Number analyzed (Participants) | 3 | 12 | 13
score on a scale | 9.3 (3.1) | 14.5 (8.2) | 13.0 (8.4)

3. Secondary Outcome: Quality of Life - General Health Score
Description: Assessed by the World Health Organization Quality of Life measure, measure reflects overall health as an indicator of quality of life. The scale range of possible scores is 2-10, with higher scores reflected better outcome (i.e., better general health).
Time Frame: Week 12
Population: Due to partial missing data, not all participants are included in this analysis. Specifically 2 people are missing from the RCT:I-CBT arm and 3 from the RCT IDC arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | I-CBT Feasibility Pilot | RCT: I-CBT | RCT IDC
Number analyzed (Participants) | 3 | 11 | 10
score on a scale | 5.7 (2.9) | 5.9 (1.2) | 6.8 (1.5)

4. Secondary Outcome: Non-opioid Substance Use
Description: Days of other substance use in the past 30 days
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | I-CBT Feasibility Pilot | RCT: I-CBT | RCT IDC
Number analyzed (Participants) | 3 | 11 | 10
days | 9.3 (16.2) | 4.8 (9.3) | 7.8 (13.6)

5. Secondary Outcome: Functional Impairment
Description: Assessed by the Addiction Severity Index (ASI) Drug Severity Score, this score reflects the severity of functional impairment due to drug use. Higher scores reflect more interference (worse outcome) and the range of scores is 0-1.
Time Frame: Week 12
Population: Due to partial missing data, 2 participants are missing from the RCT ICBT arm and 3 from the RCT IDC arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | I-CBT Feasibility Pilot | RCT: I-CBT | RCT IDC
Number analyzed (Participants) | 3 | 11 | 10
score on a scale | .15 (.14) | .10 (.10) | .07 (.05)

6. Other Pre Specified Outcome: Patient Satisfaction
Description: Assessed by the Client Satisfaction Questionnaire (CSQ), this measure assesses patient satisfaction with treatment. Higher scores reflect higher satisfaction (better outcome). The scores range from 8-32.
Time Frame: Week 12
Population: Due to partial missing data, 2 participants are missing from the RCT ICBT arm and 2 from the RCT IDC arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | I-CBT Feasibility Pilot | RCT: I-CBT | RCT IDC
Number analyzed (Participants) | 3 | 11 | 11
score on a scale | 32 (0) | 26.9 (4.8) | 29.4 (3.2)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | I-CBT Feasibility Pilot | RCT I-CBT | RCT IDC
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/5 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT02252068/Prot_SAP_000.pdf